CLINICAL TRIAL: NCT02724852
Title: Seroprevalence of Antibodies to Measles, Mumps, and Rubella, and Serologic Responses After Vaccination Among Human Immunodeficiency Virus (HIV)-1 Infected Adults in Northern Thailand
Brief Title: MMR Vaccination Among HIV-infected Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Romanee Chaiwarith, Associate Professor, Chiang Mai University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Research ID: 268
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: HIV
Keywords: MMR; vaccination; HIV; Serologic response
MeSH Terms: interventions — Measles-Mumps-Rubella Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV-infected adults (Active Comparator): Two-hundreds and forty-nine HIV-infected participants received a single dose of MMR vaccine (GlaxoSmithKline Biologicals) at deltoid region.
  Interventions were a single dose of 0.5 ml of MMR vaccine. Each 0.5 ml of vaccine contained at least 1000 TCID50 of Schwarz measles strain, at least 1000 TCID50 of RIT 4385 mumps, and at least 1000 TCID50 of Wistar RA 27/3 rubella strains.
  Interventions: Biological: 0.5 ml of MMR vaccine
- HIV-uninfected adults (Experimental): Forty-six HIV-uninfected participants received a single dose of MMR vaccine (GlaxoSmithKline Biologic) at deltoid region.
  Interventions were a single dose of 0.5 ml of MMR vaccine. Each 0.5 ml of vaccine contained at least 1000 TCID50 of Schwarz measles strain, at least 1000 TCID50 of RIT 4385 mumps, and at least 1000 TCID50 of Wistar RA 27/3 rubella strains.
  Interventions: Biological: 0.5 ml of MMR vaccine

INTERVENTIONS:
Biological: 0.5 ml of MMR vaccine — Participants in each arm received the same vaccine, a 0.5 ml of MMR vaccine at deltoid region

SUMMARY:
This is a prevalence study of protective antibodies to measles, mumps, and rubella (MMR) in HIV-infected adults and HIV-uninfected controls. MMR vaccination were provided to both groups who had no protective antibodies to at least one of the three viruses.

DETAILED DESCRIPTION:
From July to August 2011, 500 HIV-infected and 132 HIV-uninfected participants those met the eligibility criteria were enrolled and tested for protective antibodies to measles, mumps, and rubella.

All participants who had no protective antibody to at least one of the three viruses were recruited to vaccinate for MMR vaccine. Between June to September 2012, 249 HIV-infected and 46 HIV-uninfected adults were vaccinated. Antibodies to MMR were measured at week 8-12, and week 48 after vaccination, which were completed in August 2013. The results were ready for analysis in March 2014.

ELIGIBILITY:
Inclusion Criteria:

For HIV-infected participants, inclusions criteria were

1. 20-59 years old, ability to provide informed consent
2. receiving cART
3. CD4 cell count ≥200 cell/mm3 within 6 months before enrollment
4. plasma HIV-1 RNA <50 copies/mL, and 5) ability to provide informed consent.

Exclusion Criteria:

For both groups

1. pregnancy or lactating
2. receiving cancer treatment, organ transplantation, ≥0.5 mg/kg/day of prednisolone or equivalent, or immunomodulating treatment
3. impaired renal function (creatinine clearance <30 mL/min)
4. impaired liver function as defined by Child-Pugh C.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 632 (Actual)
Dates: Start 2011-07; Primary Completion 2013-09 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with protective antibodies to measles, mumps, and rubella | Baseline
  Comparison of proportions of participants who had protective antibodies to measles between HIV-infected participants and HIV-uninfected participants

SECONDARY OUTCOMES:
Proportion of participants with protective antibodies to measles, mumps, and rubella | 8-12 weeks after a single dose of MMR vaccination
  Comparison of proportion of participants who had protective antibodies to measles, mumps, and rubella between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
Proportion of participants with protective antibodies to measles, mumps, and rubella | 48 weeks after a single dose of MMR vaccination
  Comparison of proportion of participants who had protective antibodies to measles, mumps, and rubella between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-measles IgG level | 8-12 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-measles IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-measles IgG level | 48 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-measles IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-mumps IgG titers | 8-12 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-mumps IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-mumps IgG titers | 48 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-mumps IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-rubella IgG level | 8-12 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-rubella IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
The geometric means of anti-rubella IgG level | 48 weeks after a single dose of MMR vaccination
  Comparison of the geometric means of anti-rubella IgG level between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses
Proportion of participants who had adverse effects from vaccination | 72 hours after MMR vaccination
  Comparison of proportion of participants who had adverse effects from MMR vaccination between HIV-infected participants and HIV-uninfected participants in those without protective antibody to at least one of the three viruses

CONTACTS AND LOCATIONS:
Overall Officials: Romanee Chaiwarith, MD, Principal Investigator — Chiang Mai University
Locations (1):
- Maharaj Nakorn Chiang Mai Hospital, Department of Medicine, Chiang Mai University, Muang, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaiwarith R, Praparattanapan J, Nuket K, Kotarathitithum W, Supparatpinyo K. Seroprevalence of antibodies to measles, mumps, and rubella, and serologic responses after vaccination among human immunodeficiency virus (HIV)-1 infected adults in Northern Thailand. BMC Infect Dis. 2016 Apr 30;16:190. doi: 10.1186/s12879-016-1499-x. PMID 27138005